CLINICAL TRIAL: NCT05047211
Title: A Feasibility Trial of Intravenous Iron vs. Oral Iron Supplementation for the Treatment of Postpartum Anemia (IVIRONMAN)
Brief Title: Intravenous Iron vs. Oral Iron Supplementation for Postpartum Anemia
Acronym: IVIRONMAN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21-0127
Record Dates: First submitted 2021-09-07; First posted 2021-09-17 (Actual); Results first posted 2023-08-29 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Anemia, Iron Deficiency; Delivery Complication
Keywords: Postpartum, iron deficiency anemia, intravenous iron
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — ferrous sulfate; Iron-Dextran Complex

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blinded placebo controlled clinical trial. We will be using intravenous and oral placebos for each interventions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral Iron group (Active Comparator): Ferrous sulfate 325 mg (65 mg elemental iron) by mouth for a total of 6 weeks three times daily.
  Intravenous placebo in sodium chloride 0.9% 500mL IV infusion will be given before discharge home over 1 hour preceded by placebo test dose IV infusion of 100mL 0.9% sodium chloride.
  Interventions: Drug: Ferrous sulfate
- IV Iron group (Experimental): Low molecular weight iron dextran (infed) 1000mg in sodium chloride 0.9% 500mL IV infusion over 1 hour preceded by test dose 25 mg IV low molecular weight iron dextran infusion in 100mL 0.9% sodium chloride.
  Oral placebo will be given by mouth for a total of 6 weeks TID.
  Interventions: Drug: Iron dextran

INTERVENTIONS:
Drug: Ferrous sulfate — one tablet 325 milligrams three times a day
  Arms: Oral Iron group
Drug: Iron dextran — 1000 mg intravenous infusion
  Arms: IV Iron group

SUMMARY:
This trial will be a comparative pragmatic open label feasibility randomized controlled trial of oral daily versus IV iron in anemic postpartum patients.

Two randomly assigned groups will be compared during the postpartum period:

1. Oral Iron group: Ferrous sulfate 325 mg (65 mg elemental iron) by mouth for a total of 6 weeks TID.

   IV placebo in sodium chloride 0.9% 500mL IV infusion will be given before discharge home over 1 hour preceded by placebo test dose IV infusion of 100mL 0.9% sodium chloride.
2. IV Iron group: Low molecular weight iron dextran (infed) 1000mg in sodium chloride 0.9% 500mL IV infusion over 1 hour preceded by test dose 25 mg IV low molecular weight iron dextran infusion in 100mL 0.9% sodium chloride.

2.1 Oral placebo will be given by mouth for a total of 6 weeks TID.

ELIGIBILITY:
Inclusion Criteria:

* Delivery at our institution
* Hemoglobin below 9 g/dl in postpartum day 1
* Singleton gestation

Exclusion Criteria:

* Diagnosis of malabsorptive disorder or history of gastric bypass procedure
* Known diagnosis of anemia other than iron deficiency (thalassemia, macrocytic anemia, sickle cell, etc.)
* Significant cardiovascular disease, including but not limited to myocardial infarction or unstable angina within 6 months prior to study inclusion or current history of NYHA Class III or IV congestive heart failure
* Patient has received blood transfusion or there is a plan to transfuse
* Lactose intolerance

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participant eligibility is based on self-representation of gender identity.
Enrollment: 40 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-04-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ashley Salazar, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saad AF, Stepanek R, Kothmann M, Wilson-Jimenez M, McCoy L, Aguillon B, Salazar A, Saade GR. Intravenous Iron Compared With Oral Iron Supplementation for the Treatment of Postpartum Anemia: A Randomized Controlled Trial. Obstet Gynecol. 2023 Jun 1;141(6):1052-1055. doi: 10.1097/AOG.0000000000005143. Epub 2023 May 3. PMID 37486650

RESULTS

PARTICIPANT FLOW:
Groups:
- Oral Iron Group: Ferrous sulfate 325 mg (65 mg elemental iron) by mouth for a total of 6 weeks three times daily.
  Intravenous placebo in sodium chloride 0.9% 500mL IV infusion will be given before discharge home over 1 hour preceded by placebo test dose IV infusion of 100mL 0.9% sodium chloride.
  Ferrous sulfate: one tablet 325 milligrams three times a day
- IV Iron Group: Low molecular weight iron dextran (infed) 1000mg in sodium chloride 0.9% 500mL IV infusion over 1 hour preceded by test dose 25 mg IV low molecular weight iron dextran infusion in 100mL 0.9% sodium chloride.
  Oral placebo will be given by mouth for a total of 6 weeks TID.
  Iron dextran: 1000 mg intravenous infusion
Period: Overall Study
Arm/Group | Oral Iron Group | IV Iron Group
Started | 20 | 20
Completed | 12 | 15
Not Completed | 8 | 5
Not completed — Lost to Follow-up | 8 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Iron Group | IV Iron Group | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Median (Full Range); unit: years] | 24 [18 to 40] | 31 [18 to 42] | 27 [18 to 42]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin Level
Description: hemoglobin in grams per deciliters
Time Frame: 6 weeks after delivery
Measure: Median (Full Range); unit: grams/deciliters
Arm/Group | Oral Iron Group | IV Iron Group
Number analyzed (Participants) | 12 | 15
grams/deciliters | 12 [10 to 13] | 12 [11 to 14]

2. Secondary Outcome: Number of Participants With Nausea or Vomiting
Description: feeling sick to vomit or vomit
Time Frame: up to 6 weeks after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Iron Group | IV Iron Group
Number analyzed (Participants) | 19 | 17
Participants | 0 | 0

3. Secondary Outcome: Myalgia
Description: Generalized muscle pain
Time Frame: up to 6 weeks after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Iron Group | IV Iron Group
Number analyzed (Participants) | 19 | 17
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: up to 6 weeks
Arm/Group | Oral Iron Group | IV Iron Group
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-10): https://cdn.clinicaltrials.gov/large-docs/11/NCT05047211/Prot_SAP_001.pdf